CLINICAL TRIAL: NCT01926340
Title: The Impact of Early Medication Discontinuation on Long-term Clinical Outcome in First Episode Psychosis
Brief Title: Early Medication Discontinuation and Long-term Clinical Outcome in FEP
Acronym: FEP
Status: Completed | Type: Observational
Sponsor: Professor Eric Y.H. Chen (Other)
Collaborators: Research Grants Council, Hong Kong (Other); AstraZeneca (Industry); Food and Health Bureau, Hong Kong (Other Government); University of British Columbia (Other)
Responsible Party: Sponsor-Investigator, Professor Eric Y.H. Chen, Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Other Study IDs: RPS FU study
Record Dates: First submitted 2013-07-02; First posted 2013-08-20 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Early maintenance treatment group: Drug (quetiapine, 400mg/d) during the 12-month randomized phase of the study
- Early discontinuation group: Drug (placebo) during the 12-month randomized phase of the study

SUMMARY:
The study aims to examine the relationship between early maintenance therapy decisions in first episode psychosis, and the subsequent long-term clinical outcome at 9-10 years by comparing a group of patients who were randomized to discontinue (placebo) or continue medication (quetiapine) in the early stage of their psychotic disorders.

DETAILED DESCRIPTION:
Design: This is a follow up or extension to the double-blind randomized placebo-controlled 12-month study (Chen et al., BMJ 2010;341:C4024-4). At any point during the 12-month study, patients who had relapsed or discontinued would stop the study medication (quetiapine or placebo) and that would be the end point of the randomized phase of the study. After completion of the randomized phase, patients will receive clinical guideline-based, open-label treatment. Trained research assistants will approach patients at their upcoming out-patient consultations to introduce the follow-up study and to obtain their written informed consent.

Data analysis plan & handling of missing outcome data: Statistical analyses will be carried out according to the intention-to-treat principle. The primary outcome measure of the long-term clinical outcomes (suicide, clozapine treatment, persistent positive symptoms) between the groups randomized to early treatment discontinuation (placebo) or maintenance treatment (quetiapine) will be compared using risk ratios [RR] and 95% confidence intervals [CI].

For all patients, long-term outcome assessments will include longitudinal chart review over the follow-up period indicating suicide or clozapine treatment. Positive symptom will be assessed at the 10-year face-to-face interview, or in the situations where this data is not available, will be based on the last positive symptom assessment from the randomized study. We will assess the possible effect of this approach by conducting sensitivity analyses, namely re-classifying patients with missing end-point interviews as either all good outcome, or all poor outcome. A mediation analysis will also carried out to examine whether the effects of the intervention on long-term outcome are linked to relapse during the randomized phase.

The secondary outcome measures of social and occupational functioning will be analysed using RR or independent t-tests. Standardized mortality ratios (SMRs) based on age-sex population mortality rate and age-sex suicide rate will also be calculated.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of schizophrenia or non-affective psychosis (schizophreniform disorder, schizoaffective disorder, brief psychotic disorder, or psychosis not otherwise specified) (DSM-IV)
* Aged 18 to 65 years
* Had been treated with antipsychotic drugs for at least 12 months
* No history of relapse or exacerbation or had to be asymptomatic (free of positive symptoms of psychosis) at study entry.

Exclusion Criteria:

* A diagnosis of drug-induced psychosis
* Current treatment with clozapine, with mood stabilizing medications (lithium, valproate or carbamazepine) or with depot medication
* Had high risk of suicide or violence
* Had poor adherence to treatment (missing>50% of drug, >50% missed clinic visits, or a history of medication discontinuation)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trained research assistants will approach patients at their upcoming out-patient consultations to introduce the follow-up study and to obtain written informed consent. Those who are not active cases in the Hong Kong Hospital Authority (HA) system will be invited by letter and telephone to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Poor clinical outcome | In one month previous to the final assessment
  Define categorically as any of: persistent positive symptoms of psychosis, requirement for clozapine or death from suicide.
  Good clinical outcome: meeting none of the criteria for Poor clinical outcome (as above)

SECONDARY OUTCOMES:
Social and occupational functioning | In one month previous to the final assessment
  Define using employment status, social and occupational functioning score, and role functioning score

OTHER OUTCOMES:
Relapse | During the randomized phase of the study
  Define as recurrence of positive symptoms
Quality of life | In one month previous to the final assessment
  SF-36 physical and mental health summary scores

CONTACTS AND LOCATIONS:
Overall Officials: Eric YH Chen, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Research Site, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Hui CLM, Honer WG, Lee EHM, Chang WC, Chan SKW, Chen ESM, Pang EPF, Lui SSY, Chung DWS, Yeung WS, Ng RMK, Lo WTL, Jones PB, Sham P, Chen EYH. Long-term effects of discontinuation from antipsychotic maintenance following first-episode schizophrenia and related disorders: a 10 year follow-up of a randomised, double-blind trial. Lancet Psychiatry. 2018 May;5(5):432-442. doi: 10.1016/S2215-0366(18)30090-7. Epub 2018 Mar 15. PMID 29551618